CLINICAL TRIAL: NCT02446756
Title: Clinical Observation and MRI Influence of Acupuncture on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUMCH20150430
Record Dates: First submitted 2015-05-06; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Knee Arthritis Osteoarthritis
Keywords: Osteoarthritis; MRI; Cartilage; Acupuncture
MeSH Terms: conditions — Osteoarthritis | interventions — Acupuncture Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture group (Experimental): Acupuncture treatment was given once every other day and 20min each time for four weeks.
  Interventions: Other: acupuncture
- physiotherapy group (Active Comparator): Physiotherapy treatment was given five times a week and 30min each time for four weeks.
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: acupuncture
  Arms: acupuncture group
Other: physiotherapy
  Arms: physiotherapy group

SUMMARY:
To observe the therapeutic effect of acupuncture on osteoarthritis(OA) and its efficacy on cartilage restoration,acupuncture and physiotherapy treatment were respectively given to two random groups. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used to evaluate the motor function of knee joints, followed by magnetic resonance imaging (MRI) scanning to measure T2 values in ten cartilage sub-regions in tibiofemoral joints.

DETAILED DESCRIPTION:
To observe the therapeutic effect of acupuncture on osteoarthritis and its efficacy on cartilage restoration,one hundred knees of 50 patients with knee osteoarthritis were randomly divided into acupuncture group and physiotherapy group which were respectively received acupuncture and physiotherapy treatment for four weeks. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used to evaluate the motor function of knee joints, followed by magnetic resonance imaging (MRI) scanning to measure T2 values in ten cartilage sub-regions in tibiofemoral joints.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as knee osteoarthritis according to the OA criteria proposed by American College of Rheumatology in 1995.

Exclusion Criteria:

* Acute knee injury
* Had ever accepted therapy as hormone or injection in articulation cavity
* Had ever accepted treatment as oral medicine, physiotherapy, acupuncture or massage during the passed three months
* Had planted cardiac pacemaker or any metal matter in body
* Other severe diseases such as heart, lung, liver, kidney or cerebrum failure, tumors, gastrointestinal hemorrhage and so on
* Pregnant or lactating woman
* Anyone unable to tolerate or cooperate with treatment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
WOMAC scores | up to 24 months
T2 Values | up to 30 months